CLINICAL TRIAL: NCT07344792
Title: Physician Diagnosis of Neurologic Cases Assisted by Large Language Models: A Randomized Controlled Trial
Brief Title: Physician Diagnosis of Neurologic Cases With Large Language Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LLM-001
Record Dates: First submitted 2025-12-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neurology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLM assistance group (Experimental): Physicians are assisted by an in-house LLM and are allowed to use conventional resources. Access to any other LLMs is not permitted.
  Interventions: Other: LLM assistance
- Conventional assistance group (No Intervention): Physicians use only conventional resources and do not have access to the in-house LLM or any other LLMs at any point during the study.

INTERVENTIONS:
Other: LLM assistance — Physicians are assisted by an in-house large language model and are allowed to use conventional resources. Access to any other LLMs is not permitted.
  Arms: LLM assistance group

SUMMARY:
This study is a prospective randomized controlled trial that aims to evaluate whether large language model (LLM) assistance improves physicians' diagnostic performance compared with conventional assistance.

DETAILED DESCRIPTION:
The study population consists of licensed physicians who have completed at least two years of neurology training. Participants are randomly assigned in a 1:1 ratio to the LLM assistance group or the conventional assistance group. In the LLM assistance group, physicians are assisted by an in-house LLM and are allowed to use conventional resources (e.g., search engines, UpToDate, or clinical guidelines) before submitting a final diagnosis. Access to any other LLMs is not permitted. In the conventional assistance group, physicians use only conventional resources and do not have access to the in-house LLM or any other LLMs at any point during the study. The primary outcome is top-1 diagnostic accuracy. Secondary outcomes include top-3 diagnostic accuracy, the time required to complete each case, and physicians' diagnostic confidence.

ELIGIBILITY:
Inclusion Criteria:

* Licensed physicians who have completed at least two years of neurology training.
* Willing to participate in the study and able to provide written informed consent.

Exclusion Criteria:

* Physicians who have previously participated in the development of the in-house LLM or the construction of datasets used in this study.
* Physicians who were involved in the clinical care of patients whose cases were used to construct the case dataset for this study.
* Physicians who are known to have previously reviewed or been exposed to the specific cases used in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Top-1 diagnostic accuracy | Baseline
  Top-1 diagnosis is considered correct if the physician's final top-ranked diagnosis matches the reference diagnosis or a clinically similar diagnosis judged as equivalent by neurologists.

SECONDARY OUTCOMES:
Top-3 diagnostic accuracy | Baseline
  Top-3 diagnosis is considered correct if the reference diagnosis or a clinically similar diagnosis judged as equivalent by neurologists appears among the physician's top three final diagnoses.
Time spent on diagnosis | Baseline
  Time participants spend per case.
Diagnostic confidence | Baseline
  Physicians' diagnostic confidence will be measured using a five-point Likert scale (1=very unsure, 5=very sure).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Luhe Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Nanyang Central Hospital, Nanyang, Henan